CLINICAL TRIAL: NCT00814047
Title: The Effect of an α2-Adrenoceptor Antagonist (Yohimbine) on Dynamic Autoregulation in the Human Middle Cerebral Artery and Ophthalmic Artery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gabriele Fuchsjaeger-Mayrl, MD, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OPHT-280604
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Blood Flow Velocity; Autoregulation; Ocular Physiology
Keywords: ultrasonography
MeSH Terms: interventions — Yohimbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Yohimbine hydrochloride

SUMMARY:
Blood flow autoregulation is defined as the ability of a tissue to maintain a relatively constant flow, despite moderate alterations in perfusion pressure. Similar to the cerebral, renal, coronary and skeletal muscle circulations, the ocular vascular bed shows the property of flow autoregulation. This homeostatic mechanism allows blood supply to the eye to match metabolic demand during daily activities, such as changes in posture, or in more critical conditions.

Autoregulation has been found to be a complex phenomenon, showing heterogeneity in its site and time course of action. Since metabolic, myogenic, neurogenic and possibly endothelium-related mechanisms may be involved, several factors may vary depending on the challenging stimulus, the vessel tone, or the degree of impairment of autoregulation.

To study the dynamics of ocular autoregulation, it is necessary to introduce a step disturbance (stimulus) in ocular perfusion pressure and to record the responses of ocular blood flow continuously before and after this step disturbance. The investigators have employed a mechanical noninvasive technique to induce an ocular perfusion pressure step disturbance without drugs or changes in the concentration of vasoactive substances in the blood by using the thigh cuff technique inducing a small step decrease in ocular perfusion pressure.

With this technique the investigators could show significant differences in the time response of blood velocities in the ophthalmic and middle cerebral artery. This clearly indicates different mechanisms to be responsible for autoregulatory mechanisms distal to the vessels.

Interestingly our results indicate that in the ophthalmic artery a late vasoconstriction occurs. Many previous investigations have demonstrated that sympathetic nerve stimulation causes vasoconstriction in the ocular circulation. Accordingly, the present study tests the hypothesis that α2-adrenoceptors are involved in the dynamic regulation of blood flow in the ophthalmic and middle cerebral artery after a step decrease in perfusion pressure.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 35 years
* Non-smokers
* Normal findings in medical history and pre-study screening unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 3 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18

PRIMARY OUTCOMES:
Relation between blood pressure and local perfusion parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjäger-Mayrl, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria